CLINICAL TRIAL: NCT03086629
Title: Improving Quality of Life Through the Routine Use of the Patient Concerns Inventory for Head and Neck Cancer Patients (PCI-QoL)
Brief Title: Improving Quality of Life Through the Routine Use of the Patient Concerns Inventory for Head and Neck Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Collaborators: The Leeds Teaching Hospitals NHS Trust (Other); National Institute for Health Research, United Kingdom (Other Government); Bangor University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 16/NW/0465
Record Dates: First submitted 2016-08-01; First posted 2017-03-22 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2018-07

CONDITIONS: Cancer of Head and Neck
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCI Group (Other): Participants who are patients of consultants randomized to this group will use the PCI during clinics.
  Interventions: Other: Patient Concerns Inventory
- Non PCI Group (Other): Participants who are patients of consultants randomized to this group will not use the PCI during clinics.
  Interventions: Other: No Patient Concerns Inventory

INTERVENTIONS:
Other: Patient Concerns Inventory
  Other Names: PCI Group
  Arms: PCI Group
Other: No Patient Concerns Inventory
  Other Names: Non PCI Group
  Arms: Non PCI Group

SUMMARY:
The Patient Concerns Inventory (PCI) for head and neck cancer (HNC) patients has been developed and used largely within the confines of a single clinic setting and has not been used routinely with patients in the first year following treatment. Research so far suggests it is popular with patients, they would like to continue to use it in clinic and it is feasible. Benefits of its routine repeated use is untested, notably its impact on improving QOL and in reducing emotional distress, especially within the first year after treatment when patients are more likely to benefit from repeated use of the PCI.

The overarching aim of the proposed research is to explore whether the routine use of the PCI in review clinics during the first year following head and neck cancer treatment can improve patients quality of life.

The primary outcome is an improvement in QOL. Secondary outcomes are:

social-emotional scale, distress thermometer and health economics.

This will be a pragmatic cluster randomised control trial with consultants randomised to either 'using or 'not using' the PCI at clinic. It will involve two centres. 416 patients from at least 10 consultant clusters are required to show a clinically meaningful difference in the primary outcome.

Intervention; Patient completion of the PCI and its inclusion into the regular review clinic consultation is the 'intervention' and is compared to standard out-patient follow-up. The pre-consultation questionnaires and PCI will be used from the first post-treatment clinic (i.e. baseline) onwards for one year. Completion of all pre-consultation questionnaires and the PCI is by computer (IPAD).

DETAILED DESCRIPTION:
The Patient Concerns Inventory (PCI) for head and neck cancer (HNC) patients has been developed and used largely within the confines of a single clinic setting and has not been used routinely with patients in the first year following treatment. Research so far suggests it is popular with patients, they would like to continue to use it in clinic and it is feasible. Benefits of its routine repeated use is untested, notably its impact on improving QOL and in reducing emotional distress, especially within the first year after treatment when patients are more likely to benefit from repeated use of the PCI.

The overarching aim of the proposed research is to explore whether the routine use of the PCI in review clinics during the first year following head and neck cancer treatment can improve patients quality of life.

The primary outcome is the percentage of participants with less than good overall quality of life at the final one-year clinic as measured by the single UWQOLv4 question.

Secondary outcomes at one-year are the mean social-emotional subscale (UWQOLv4) score, Distress Thermometer (DT) score ≥4, and key health economic measures (QALY-EQ-5D-5L; CSRI).

This will be a pragmatic cluster randomised control trial with consultants randomised to either 'using or 'not using' the PCI at clinic. It will involve two centres. 416 patients recruited from 14 MFU and ENT consultants are required to show a clinically meaningful difference in the primary outcome.

Intervention: Patient completion of the PCI and its inclusion into the regular review clinic consultation is the 'intervention' and is compared to standard out-patient follow-up. The pre-consultation questionnaires and PCI will be used from the first post-treatment clinic (i.e. baseline) onwards for one year. Completion of all pre-consultation questionnaires and the PCI is by computer (IPAD).

ELIGIBILITY:
Inclusion Criteria:

* Patients with HNC
* To be treated curatively (all sites, stage of disease, treatments).

Exclusion Criteria:

* Patients treated with palliative intent
* Patients with a recurrence.
* Patients with a history of cognitive impairment, psychoses or dementia

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
UWQOL v4 QoL | Post-Treatment 1 Year Review Clinic
  The percentage of participants with less than good overall quality of life at the final one-year clinic.

SECONDARY OUTCOMES:
UWQOL v4 Questionnaire | Post-Treatment 1 Year Review Clinic
  Mean social-emotional subscale score
Distress Thermometer VAS | Post-Treatment 1 Year Review Clinic
  Score ≥4
QALY-EQ-5D-5L | Post-Treatment 1 Year Review Clinic
  Key health economics questionnaire
CSRI | 6 Month and 12 Month Post-Treatment Review Clinics
  Key health economics questionnaire

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - St Helens & Knowsley Teaching Hospitals NHS Trust, Liverpool, Merseyside
  - Aintree University Hospital NHS Foundation Trust, Liverpool, Merseyside
  - Leeds Teaching Hospitals Nhs Trust, Leeds, Yorkshire

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kanatas A, Lowe D, Rogers SN. Health-related quality of life at 3 months following head and neck cancer treatment is a key predictor of longer-term outcome and of benefit from using the patient concerns inventory. Cancer Med. 2022 Apr;11(8):1879-1890. doi: 10.1002/cam4.4558. Epub 2022 Feb 17. PMID 35178880
- [Derived] Ezeofor V', Spencer LH, Rogers SN, Kanatas A, Lowe D, Semple CJ, Hanna JR, Yeo ST, Edwards RT. An Economic Evaluation Supported by Qualitative Data About the Patient Concerns Inventory (PCI) versus Standard Treatment Pathway in the Management of Patients with Head and Neck Cancer. Pharmacoecon Open. 2022 May;6(3):389-403. doi: 10.1007/s41669-021-00320-4. Epub 2022 Jan 31. PMID 35099783
- [Derived] Rogers SN, Lowe D, Lowies C, Yeo ST, Allmark C, Mcavery D, Humphris GM, Flavel R, Semple C, Thomas SJ, Kanatas A. Improving quality of life through the routine use of the patient concerns inventory for head and neck cancer patients: a cluster preference randomized controlled trial. BMC Cancer. 2018 Apr 18;18(1):444. doi: 10.1186/s12885-018-4355-0. PMID 29669529